CLINICAL TRIAL: NCT04416685
Title: A New Anatomical Classification of Portal Venous Involvement in Locally Advanced Pancreatic Cancer to Predict the Surgical Difficulty
Brief Title: A New Anatomical Classification of Portal Vein Location of Pancreas Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pinar Yazici, Assoc Prof, Sisli Hamidiye Etfal Training and Research Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PVR-2019
Record Dates: First submitted 2020-05-31; First posted 2020-06-04 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-04

CONDITIONS: Pancreatic Neoplasm Malignant Head Primary
Keywords: pancreas tumors
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Mastectomy, Segmental

STUDY DESIGN:
Intervention Model Description: Anatomical classification was established based on the relationship between portal confluence (PC) and tumor location . Those tumors located superior to the PC were classified as Level I, whereas tumors on the confluence inferiorly located to PC were classified as Level II and Level III.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Level 1 (Other): Those tumors located superior to the portal confluence were classified as Level I,
  Interventions: Procedure: primary repair; Procedure: segmental resection
- Level II (Other): those tumors located on the confluence (involving the confluence) located on the portal confluence
  Interventions: Procedure: primary repair; Procedure: segmental resection
- Level III (Other): those tumors located inferior to the portal confluence
  Interventions: Procedure: segmental resection; Procedure: graft reconstruction

INTERVENTIONS:
Procedure: primary repair — For Level I-II tumors, in case of segmental resection of PV/SMV, the reconstruction was performed by an end-to-end anastomosis either by direct suture (for defect under 2 cm) or by using an interposition venous or prosthetic graft. For this purpose, autologous grafting we used internal jugular vein and cadaveric iliac vein and alternatively, synthetic PTFE graft was also used.
  Arms: Level 1; Level II
Procedure: segmental resection — For Level I-II tumors, in case of segmental resection of PV/SMV, the reconstruction was performed by an end-to-end anastomosis either by direct suture (for defect under 2 cm) or by using an interposition venous or prosthetic graft. For this purpose, autologous grafting we used internal jugular vein and cadaveric iliac vein and alternatively, synthetic PTFE graft was also used.
  Other Names: primary repair
Procedure: graft reconstruction — Regarding Level III tumors, complete resection of the tumor was done either by tangential excision or by partial venous excision and subsequent reconstruction. To maintain a secure anastomosis, the mesenteric root was mobilized completely or/and splenic vein was divided.
  Other Names: segmental resection
  Arms: Level III

SUMMARY:
In this retrospective study, we recorded the location of pancreatic tumors and relation/proximity to the portal vein. The surgical difficulty and requirement of additional interventions were also evaluated.

DETAILED DESCRIPTION:
Between May 2014 and October 2018, all patients who underwent PD procedure were retrospectively reviewed. This retrospective cohort study identified all consecutive patients with T3 (stage IIA to III) adenocarcinoma of the head of the pancreas, who underwent concomitant venous (PV/SMV) resection. Those patients with locally advanced tumors that were not responded to neoadjuvant therapy were excluded. The local ethical committee was approved this study.

Data collection included demographical features, tumor characteristics including the PV level of the tumor considering computed tomography results, neoadjuvant therapy, surgical data, hospital stay, morbidity and mortality.

Anatomical classification was established based on the relationship between portal confluence (PC) and tumor location (Figure I). Those tumors located superior to the PC were classified as Level I, whereas tumors on the confluence inferiorly located to PC were classified as Level II and Level III.

ELIGIBILITY:
Inclusion Criteria:

* This retrospective cohort study identified all consecutive patients with T3 (stage IIA to III) adenocarcinoma of the head of the pancreas, who underwent concomitant venous (PV/SMV) resection.

Exclusion Criteria:

* Those patients with locally advanced tumors that were not responded to neoadjuvant therapy were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
peri-operative or postoperative complication | up to one month
  surgical complications observed during both operative and postoperative period

SECONDARY OUTCOMES:
hospital stay | up to one month
  the time between the day of surgery and hospital discharge

OTHER OUTCOMES:
in hospital mortality | up to two months
  any mortality after/during surgery in the initial hospital stay

IPD SHARING:
Plan to Share IPD: Undecided
any question about details can be shared via e-mail privately.